CLINICAL TRIAL: NCT04247893
Title: Incorporation of Photobiomodulation Therapy in an Exercise Program With Blood Flow Restriction for Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Clinical Professor., University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20123719.1.0000.5511
Record Dates: First submitted 2020-01-27; First posted 2020-01-30 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Osteoarthritis, Knee; Physical Therapy Modalities
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Blood Flow Restriction Therapy; Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Exercises with blood flow restriction (Active Comparator): Exercise: 10 minutes of heating on a treadmill without changing the inclination and adopting a standardized speed; Supine bridge, Supine unilateral bridge, Flexion of the hip with the knee extended, Knee extension, volunteer in sedation; Prone knee flexion; Squat on the wall associated with isometric contraction; Abduction of the hip, lateral rotation and knee extension in lateral decubitus associated with isometric contraction; Abduction, lateral rotation of the hip, slight knee and hip flexion performing abduction with the feet together: associated with isometric contraction; Abduction of the hip in orthostatic associated with isometric contraction.Device: The blood flow restriction in mmHg will be performed using a vascular occlusion training manometer, positioned in the thigh inguinal region and inflated to the point where the auscultatory pulse of the tibial artery is interrupted.
  Interventions: Device: blood flow restriction
- Exercises with blood flow restriction + photobiomodulation (Experimental): Exercise: 10 minutes of heating on a treadmill without changing the inclination and adopting a standardized speed; Supine bridge, Supine unilateral bridge, Flexion of the hip with the knee extended, Knee extension, volunteer in sedation; Prone knee flexion; Squat on the wall associated with isometric contraction; Abduction of the hip, lateral rotation and knee extension in lateral decubitus associated with isometric contraction; Abduction, lateral rotation of the hip, slight knee and hip flexion performing abduction with the feet together: associated with isometric contraction; Abduction of the hip in orthostatic associated with isometric contraction.Devices: The blood flow restriction in mmHg will be performed using a vascular occlusion training manometer, positioned in the thigh inguinal region and inflated to the point where the auscultatory pulse of the tibial artery is interrupted.Photobiomodulation a mesh composed of multiple diodes containing 50 Infrared LEDs.
  Interventions: Device: blood flow restriction; Device: Photobiomodulation
- Blood flow restriction exercises + placebo photobiomodulation (Placebo Comparator): Exercise: 10 minutes of heating on a treadmill without changing the inclination and adopting a standardized speed; Supine bridge, Supine unilateral bridge, Flexion of the hip with the knee extended, Knee extension, volunteer in sedation; Prone knee flexion; Squat on the wall associated with isometric contraction; Abduction of the hip, lateral rotation and knee extension in lateral decubitus associated with isometric contraction; Abduction, lateral rotation of the hip, slight knee and hip flexion performing abduction with the feet together: associated with isometric contraction; Abduction of the hip in orthostatic associated with isometric contraction.Devices: The blood flow restriction in mmHg will be performed using a vascular occlusion training manometer, positioned in the thigh inguinal region and inflated to the point where the auscultatory pulse of the tibial artery is interrupted. Photobiomodulation turned off with a mesh composed of multiple diodes containing 50 Infrared LEDs.
  Interventions: Device: blood flow restriction; Device: Placebo photobiomodulation

INTERVENTIONS:
Device: blood flow restriction — Occlusion training is an exercise approach whereby resistance exercise or aerobic exercise is performed whilst an occlusion cuff is applied to proximal aspect of the muscle.
Device: Photobiomodulation — Photobiomodulation therapy is defined as the utilization of non-ionizing electromagnetic energy to trigger photochemical changes within cellular structures that are receptive to photons.
  Arms: Exercises with blood flow restriction + photobiomodulation
Device: Placebo photobiomodulation — Placebo photobiomodulation - photobiomodulation device turned off.
  Arms: Blood flow restriction exercises + placebo photobiomodulation

SUMMARY:
Knee osteoarthritis (OA) is one of the most common musculoskeletal disorders in the world. The aim of this project is to evaluate the additional effect of photobiomodulation therapy on the quadriceps muscle and knee joint in a blood flow restriction exercise program for individuals with knee OA. To this end, volunteers will be selected at random, aged between 40 and 65 years with pain in one knee, at least in the last 6 months, diagnosed with unilateral knee OA based on the criteria established by the American College of Rheumatology and radiographic confirmation for grades 2 or 3 of the Kellgren-Lawrence Classification, will be randomized into the following groups: (Exercises with blood flow restriction, n = 20), (Exercises with blood flow restriction + photobiomodulation, n = 20) and Exercises with blood flow restriction + placebo photobiomodulation (n = 20). 12 consecutive weeks of treatment will be carried out, with the volunteers being evaluated before and after, using the following instruments: The Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC), sit and stand test, Timed up and Go (TUG), numerical scale pain assessment (END), pain-to-pressure threshold (LDP), skin temperature: quadriceps musculature, knee joint and maximum voluntary isometric contraction (MVIC) of the muscles: quadriceps, middle gluteus. For data analysis, normality test will be used to verify the data distribution and statistical test consistent with the appropriate comparisons within and between groups, thus, two factors are considered in the comparisons, time and group. A significance level of 5% will be adopted.

ELIGIBILITY:
Inclusion Criteria:

* knee pain to at least six months and minimum of 4 points in pain scale
* diagnosis of unilateral knee OA based on criteria established by the American College of Rheumatology and radiographic confirmation for grades 2 or 3 of the Kellgren-Lawrence Classification.

Exclusion Criteria:

* Score on the numerical visual analog of knee pain less than 1 or greater than 8;
* knee trauma;
* Cognitive impairment;
* Psychological disorder;
* Neurological disorder (sensory or motor);
* Cancer;
* Diabetes any acute adverse health condition;
* Signs of hip OA;
* Sings cardiopulmonary disease that could prevent exercise and use of a walking assist device.
* Have undergone any form of treatment involving: physiotherapy, intra-articular corticosteroids, anti-inflammatories or chondroprotectors in the last year.
* If the size of the circumference of the thigh and knee does not allow the proper positioning of the photobiomodulation mesh.

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — As it is a disease more prevalent in women than men and more, understanding the variability in strength and muscle mass, we decided to include only female volunteers.
Enrollment: 60 (Estimated)
Dates: Start 2020-11 (Estimated); Primary Completion 2020-11 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Functional pain | Change from Baseline in The Western Ontario and McMaster Universities Arthritis Index at 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis.
Stiffness | Time Frame: Change from Baseline in The Western Ontario and McMaster Universities Arthritis Index at 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis.
Physical functional | Change from Baseline in The Western Ontario and McMaster Universities Arthritis Index at 12 weeks
  The Western Ontario and McMaster Universities Arthritis Index (WOMAC) is widely used in the evaluation Knee Osteoarthritis.

SECONDARY OUTCOMES:
Intensity of pain | Change from Baseline in The Numerical rating pain scale at 12 weeks
  The Numerical rating pain scale, a simple, easily administered scale evaluates the perceived intensity of pain, using an 11-point scale from 0, representing 'no pain', to 10, which is the 'worst possible pain'.
Functional capacity for sitting and standing | Change from Baseline in The Functional capacity for sitting and standing at 12 weeks
  sitting-rising test
Level of pressure pain | Change from Baseline in ThePressure Pain Threshold at 12 weeks
  Pressure Pain Threshold in the knee with algometer dynamometer.
Muscle skin temperature | Change from Baseline in the muscle skin temperature at 12 weeks
  Infrared thermography, thermal imaging. Thermography uses a type of infrared technology that detects and records temperature changes on the surface of the ski.
Maximum voluntary isometric contraction | Change from Baseline in the Maximum voluntary isometric contraction at 12 weeks
  A portable dynamometer will be used to assess muscle contraction.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided